CLINICAL TRIAL: NCT04308447
Title: Ablelite Pediatric Device Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AbiliTech Medical Inc. (Industry)
Collaborators: Gillette Children's Specialty Healthcare (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR610003-100; 2R44HD089789-02 (NIH)
Record Dates: First submitted 2020-02-22; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Muscular Dystrophies
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- AbleLite (Experimental): The AbleLite device is a passively powered orthotic device designed to support and assist the arms of patients with neuromuscular weakness for activities of daily living.
  Interventions: Device: AbleLite

INTERVENTIONS:
Device: AbleLite — The AbleLite device is a passively powered orthotic device designed to support and assist the arms of patients with neuromuscular weakness for activities of daily living.

SUMMARY:
The primary objective of the AbleLite early feasibility study is to evaluate the function of the upper limbs of participants diagnosed with neuromuscular disorders as children, with and without use of the Abilitech AbleLite device in the clinic and home environments. Functional outcomes will include documenting active range of motion and the ability to perform activities of daily living (ADLs) using the standardized Canadian Occupational Performance Measure (COPM) and the Role Evaluation of Activities of Life (REAL) assessments. Secondary objectives are to assess the safety record and report on adverse events (AEs) and parameters related to device usage, including device usage time and the time required to don/doff the device.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 9 and 18 years of age, with pediatric onset of neuromuscular conditions that cause quadriparesis
2. MMT score of 1-3 in the elbow, wrist and hands, and an MMT score of 2- to 3 in the shoulder
3. Ability of subject to raise their forearm off of their lap or laptray
4. Willingness to comply and participate with the study protocol and attend the study sessions
5. Ability to communicate verbally and respond to questions and commands
6. Ability to provide informed consent
7. Selected for participation based on investigator discretion

Exclusion Criteria:

1. Use of ventilator
2. Open wounds or chronic pressure sores on upper extremities, neck, back or torso
3. Significantly unstable upper extremity joints
4. Unhealed bone fractures in the upper extremities
5. Active rotator cuff tear, grade 2 or 3
6. Surgical fixations limiting full passive range of motion
7. Uncontrolled upper-limb spasticity that significantly limits normal range of motion
8. Uncontrollable pain in the neck, shoulders or upper limbs
9. Ability to fully raise both hands simultaneously above their head with ease
10. Lack passive shoulder abduction of 120 degrees
11. Lack 90 degrees of passive elbow extension
12. Unable to follow instructions
13. Exhibit significant behavioral problems
14. Inability to provide consent

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Change from Baseline before device intervention (30 days), and after device intervention (60 days)
  The Canadian Occupational Performance Measure is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time.
Roll Evaluation of Activities of Life (REAL) assessment | Change from Baseline before device intervention (30 days), and after device intervention (60 days)
  The REAL is an instrument to help professionals assess a child's ability to care for themselves at home, at school and in the community.

IPD SHARING:
Plan to Share IPD: No